CLINICAL TRIAL: NCT01923363
Title: Pharmacokinetics and Pharmacodynamics of High-Dose Piperacillin/Tazobactam in Obese Patients
Brief Title: PK/PD of High Dose Pip/Tazo in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Steven Forland, Clinical Pharmacy Specialist - Infectious Diseases, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5130259
Record Dates: First submitted 2013-08-08; First posted 2013-08-15 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: pharmacokinetics; obesity; piperacillin-tazobactam combination product; pharmacodynamics; piperacillin/tazobactam
MeSH Terms: conditions — Obesity | interventions — Piperacillin; Tazobactam; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard Dose to High Dose Piperacillin/Tazobactam (Experimental): Patients will receive a standard dose of piperacillin/tazobactam, then will have subsequent pharmacokinetic analyses on the blood concentrations drawn while on standard dose. Then, they will be switched to higher dose, with subsequent pharmacokinetic analyses performed on those blood concentrations while on higher dose. These pharmacokinetics of each dosing regimen will be compared.
  Interventions: Drug: Piperacillin/Tazobactam Standard Dose to High Dose

INTERVENTIONS:
Drug: Piperacillin/Tazobactam Standard Dose to High Dose — Patients will receive a standard dose of piperacillin/tazobactam, then will have subsequent pharmacokinetic analyses on the blood concentrations drawn while on standard dose. Patients will be switched to higher dose after receiving the standard dose, with subsequent pharmacokinetic analyses performed on those blood concentrations while on higher dose. These pharmacokinetics of each dosing regimen will be compared.
  Other Names: Zosyn

SUMMARY:
Worldwide rates of obesity have doubled in the last 30 years, and obesity has been associated as a risk factor for hospital-acquired infections and increased occurrence of death in critically-ill patients. Piperacillin/tazobactam is a commonly prescribed antibiotic for critically ill patients with an infection, however, limited information exists for dosing this drug in obese patients. In these limited reports, standard doses of piperacillin/tazobactam given to the small number of obese patients resulted in lower blood concentrations, which could lead to inadequate killing of bacteria. The purpose of this study is to compare blood concentrations from standard piperacillin/tazobactam dosing compared to higher dosing regimens in obese patients. This study will also include information on the safety and tolerability of the higher dose regimens. The study investigators believe that the higher dosing regimen will produce adequate blood levels in obese patients and will not add any more risk of harm to obese patients receiving this higher dose.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 30 kg/m2
* Weight at least 105 kg
* Age 18-89 years of age
* Prescribed piperacillin/tazobactam at standard doses for suspected or confirmed infection(s)
* English or Spanish speaking
* Central line access

Exclusion Criteria:

* Do not meet specified inclusion criteria
* Hepatic impairment classified by Child-Pugh Class B or greater
* Documented pre-existing seizure disorder
* Documented pre-existing hematologic disorder
* Pregnancy
* Documented allergy or contraindication to beta-lactams or tazobactam

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2016-01-23 (Actual); Study Completion 2016-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Forland, PharmD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veillette JJ, Winans SA, Maskiewicz VK, Truong J, Jones RN, Forland SC. Pharmacokinetics and Pharmacodynamics of High-Dose Piperacillin-Tazobactam in Obese Patients. Eur J Drug Metab Pharmacokinet. 2021 May;46(3):385-394. doi: 10.1007/s13318-021-00677-1. Epub 2021 Mar 20. PMID 33743171

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 438 obese patients receiving P-T were screened between June 2013 and January 2016. 67 patients fit inclusion criteria - 12 chose not to participate in the study or informed consent could not be obtained; 9 were excluded due to refusal of the primary care team; 13 had P-T discontinued prior to enrollment; and 4 were included previously in the study
Groups:
- Piperacillin/Tazobactam Standard to High Dose: Patients will receive a standard dose of piperacillin/tazobactam, then will have subsequent pharmacokinetic analyses on the blood concentrations drawn while on standard dose. Then, they will be switched to higher dose, with subsequent pharmacokinetic analyses performed on those blood concentrations while on higher dose. These pharmacokinetics of each dosing regimen will be compared.
Period: Overall Study
Arm/Group | Piperacillin/Tazobactam Standard to High Dose
Started | 29
Completed | 28
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Piperacillin/Tazobactam Standard to High Dose
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] — Population: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  years
    Group 1 (CrCl >/= 80mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80mL/min) | 46 [19 to 68]
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 57 [43 to 79]
    Group 3 (CrCl < 40): number analyzed (Participants) | 5
    Group 3 (CrCl < 40) | 60 [48 to 74]
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 42 [29 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28
Body Mass Index (BMI) [Median (Full Range); unit: kilograms per sqare meter] — Population: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  kilograms per sqare meter
    Group 1 (CrCl >/= 80 mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80 mL/min) | 41 [32 to 57]
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 47 [34 to 65]
    Group 3 (CrCl < 40 mL/min): number analyzed (Participants) | 5
    Group 3 (CrCl < 40 mL/min) | 38 [33 to 50]
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 49 [40 to 55]
Weight [Median (Full Range); unit: kilograms] — Population: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  kilograms
    Group 1 (CrCl >/= 80 mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80 mL/min) | 127 [105 to 151]
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 142 [118 to 205]
    Group 3 (CrCl < 40 mL/min): number analyzed (Participants) | 5
    Group 3 (CrCl < 40 mL/min) | 121 [109 to 137]
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 136 [118 to 156]
Total Bilirubin [Median (Full Range); unit: milligrams per deciliter] — Population: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  milligrams per deciliter
    Group 1 (CrCl >/= 80 mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80 mL/min) | 0.6 [0.2 to 1.5]
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 0.8 [0.4 to 1.9]
    Group 3 (CrCl < 40 mL/min): number analyzed (Participants) | 5
    Group 3 (CrCl < 40 mL/min) | 1.3 [0.3 to 3.0]
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 0.5 [0.3 to 0.9]
ICU Status [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  Participants
    Group 1 (CrCl >/= 80 mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80 mL/min) | 6
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 7
    Group 3 (CrCl < 40 mL/min): number analyzed (Participants) | 5
    Group 3 (CrCl < 40 mL/min) | 5
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 3
Acute Physiologic Assessment and Chronic Health Evaluation (APACHE) II Score [Median (Full Range); unit: units on a scale] — The APACHE II score is calculated at the beginning of the ICU admission to help determine the patient's mortality risk for the admission
  The higher the score, the higher the risk of mortality.
  Approximated Mortality Rate by score
  0-4 = 4% 5-9 = 8% 10-14 = 15% 15-19 = 25% 20-24 = 40% 25-29 = 55% 30-34 = 75% >34 = 85% Population: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  units on a scale
    Group 1 (CrCl >/= 80 mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80 mL/min) | 15.7 [9 to 26]
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 16.6 [4 to 42]
    Group 3 (CrCl < 40 mL/min): number analyzed (Participants) | 5
    Group 3 (CrCl < 40 mL/min) | 22.8 [16 to 28]
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 26.0 [21 to 29]
Sequential Organ Failure Assessment (SOFA) Score [Median (Full Range); unit: units on a scale] — Scores can be measured on all patients admitted to the intensive care unit in order to determine level of acuity and mortality risk.
  The higher the score, the higher the mortality risk.
  Mean SOFA Score Mortality 0-1.0 = 1.2% 1.1-2.0 = 5.4% 2.1-3.0 = 20.0% 3.1-4.0 = 36.1% 4.1-5.0 = 73.1% >5.1 = 84.4% Population: Measure Analysis Population Description: Patients categorized by degree of renal function. The total number of patients is 28, divided into 4 different groups based on degree of renal insufficiency as measured by creatinine clearance (CrCl).
  units on a scale
    Group 1 (CrCl >/= 80 mL/min): number analyzed (Participants) | 12
    Group 1 (CrCl >/= 80 mL/min) | 5.8 [5 to 7]
    Group 2 (CrCl >/= 40 to < 80 mL/min): number analyzed (Participants) | 8
    Group 2 (CrCl >/= 40 to < 80 mL/min) | 7.4 [0 to 14]
    Group 3 (CrCl < 40 mL/min): number analyzed (Participants) | 5
    Group 3 (CrCl < 40 mL/min) | 9.4 [6 to 11]
    Group 4 (Hemodialysis): number analyzed (Participants) | 3
    Group 4 (Hemodialysis) | 9.3 [7 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Serum Maximum Concentrations for Piperacillin
Description: Pharmacokinetic parameters for piperacillin of maximum serum concentration (Cmax) will be measured in both standard dosing and high dosing.
Time Frame: 0, 1, 3, and 6 hours post-dose
Population: The # of participants in the rows below will be double the overall participant number because each patient had two different dosing regimens of pip/tazo In Group 3, 4.5g group N = 5 represents low and high dose - 2 patients receiving 4.5g upon enrollment and increased to 6.75g; 3 patients were receiving either 2.25g or 3.375g and increased to 4.5g
Measure: Mean (Full Range); unit: milligrams per liter
Arm/Group | Standard Dose to High Dose Piperacillin/Tazobactam
Number analyzed (Participants) | 28
milligrams per liter
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams: number analyzed (Participants) | 7
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams | 136 [107 to 179]
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams | 190 [149 to 247]
  Group 1 (CrCl > 80 mL/min) on 6.75 grams: number analyzed (Participants) | 9
  Group 1 (CrCl > 80 mL/min) on 6.75 grams | 237 [96.4 to 368]
  Group 1 (CrCl >/= 80 mL/min) on 9 grams: number analyzed (Participants) | 3
  Group 1 (CrCl >/= 80 mL/min) on 9 grams | 332 [283 to 417]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 3.375 gram: number analyzed (Participants) | 6
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 3.375 gram | 144 [99.1 to 184]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 4.5 grams: number analyzed (Participants) | 2
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 4.5 grams | 214 [211 to 215]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 6.75 grams: number analyzed (Participants) | 7
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 6.75 grams | 244 [172 to 350]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 9 grams: number analyzed (Participants) | 1
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 9 grams | 191 [191 to 191]
  Group 3 (CrCl < 40 mL/min) on 2.25 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40 mL/min) on 2.25 grams | 176 [94.6 to 258]
  Group 3 (CrCl < 40 mL/min) on 3.375 grams: number analyzed (Participants) | 1
  Group 3 (CrCl < 40 mL/min) on 3.375 grams | 296 [296 to 296]
  Group 3 (CrCl < 40 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 3 (CrCl < 40 mL/min) on 4.5 grams | 265 [163 to 327]
  Group 3 (CrCl < 40 mL/min) on 6.75 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40 mL/min) on 6.75 grams | 299 [287 to 312]
  Group 4 (HD) on 2.25 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 2.25 grams | 158 [142 to 173]
  Group 4 (HD) on 3.375 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 3.375 grams | 223 [223 to 223]
  Group 4 (HD) on 4.5 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 4.5 grams | 275 [275 to 275]
  Group 4 (HD) on 6.75 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 6.75 grams | 397 [304 to 490]

2. Primary Outcome: Serum Minimum Concentrations of Piperacillin
Description: Minimum serum concentrations (Cmin) of piperacillin will be measured in both standard and high doses
Time Frame: 0, 1, 3, and 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: milligrams per liter
Arm/Group | Standard Dose to High Dose Piperacillin/Tazobactam
Number analyzed (Participants) | 28
milligrams per liter
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams: number analyzed (Participants) | 7
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams | 8.9 [0.0 to 44.1]
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams | 11.1 [1.4 to 18.2]
  Group 1 (CrCl >/= 80 mL/min) on 6.75 grams: number analyzed (Participants) | 9
  Group 1 (CrCl >/= 80 mL/min) on 6.75 grams | 27.0 [8.6 to 72.6]
  Group 1 (CrCl >/= 80 mL/min) on 9 grams: number analyzed (Participants) | 3
  Group 1 (CrCl >/= 80 mL/min) on 9 grams | 10.3 [0.57 to 29.4]
  Group 2 (CrCl >/= 40 to 80 mL/min) on 3.375 grams: number analyzed (Participants) | 6
  Group 2 (CrCl >/= 40 to 80 mL/min) on 3.375 grams | 47.4 [24.1 to 75.4]
  Group 2 (CrCl >/= 40 to 80 mL/min) on 4.5 grams: number analyzed (Participants) | 2
  Group 2 (CrCl >/= 40 to 80 mL/min) on 4.5 grams | 52.5 [49.4 to 55.6]
  Group 2 (CrCl >/= 40 to 80 mL/min) on 6.75 grams: number analyzed (Participants) | 7
  Group 2 (CrCl >/= 40 to 80 mL/min) on 6.75 grams | 72.6 [37.5 to 128]
  Group 2 (CrCl >/= 40 to 80 mL/min) on 9 grams: number analyzed (Participants) | 1
  Group 2 (CrCl >/= 40 to 80 mL/min) on 9 grams | 54.1 [54.1 to 54.1]
  Group 3 (CrCl < 40 mL/min) on 2.25 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40 mL/min) on 2.25 grams | 78.8 [14.5 to 143]
  Group 3 (CrCl < 40 mL/min) on 3.375 grams: number analyzed (Participants) | 1
  Group 3 (CrCl < 40 mL/min) on 3.375 grams | 207 [207 to 207]
  Group 3 (CrCl < 40 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 3 (CrCl < 40 mL/min) on 4.5 grams | 142 [31.1 to 223]
  Group 3 (CrCl < 40 mL/min) on 6.75 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40 mL/min) on 6.75 grams | 148 [135 to 162]
  Group 4 (HD) on 2.25 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 2.25 grams | 99 [79.6 to 118]
  Group 4 (HD) on 3.375 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 3.375 grams | 143 [143 to 143]
  Group 4 (HD) on 4.5 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 4.5 grams | 181 [181 to 181]
  Group 4 (HD) on 6.75 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 6.75 grams | 234 [193 to 274]

3. Secondary Outcome: Half-life of Piperacillin
Description: Half-life (t1/2) of piperacillin will be calculated from serum concentrations in both standard and high doses
Time Frame: 0, 1, 3, and 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Arm/Group | Standard Dose to High Dose Piperacillin/Tazobactam
Number analyzed (Participants) | 28
hours
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams: number analyzed (Participants) | 7
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams | 1.2 [0.5 to 2.7]
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams | 1.5 [0.8 to 2.4]
  Group 1 (CrCl >/= 80 mL/min) on 6.75 grams: number analyzed (Participants) | 9
  Group 1 (CrCl >/= 80 mL/min) on 6.75 grams | 1.8 [1.1 to 3.0]
  Group 1 (CrCl >/= 80 mL/min) on 9 grams: number analyzed (Participants) | 3
  Group 1 (CrCl >/= 80 mL/min) on 9 grams | 0.9 [0.6 to 1.4]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 3.375 gram: number analyzed (Participants) | 6
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 3.375 gram | 3.9 [1.9 to 6.8]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 4.5 grams: number analyzed (Participants) | 2
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 4.5 grams | 2.7 [2.6 to 2.7]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 6.75 grams: number analyzed (Participants) | 7
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 6.75 grams | 3.8 [2.2 to 9.4]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 9 grams: number analyzed (Participants) | 1
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 9 grams | 2.5 [2.5 to 2.5]
  Group 3 (CrCl < 40 mL/min) on 2.25 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40 mL/min) on 2.25 grams | 4.3 [2.0 to 6.5]
  Group 3 (CrCl < 40 mL/min) on 3.375 grams: number analyzed (Participants) | 1
  Group 3 (CrCl < 40 mL/min) on 3.375 grams | 10.7 [10.7 to 10.7]
  Group 3 (CrCl < 40 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 3 (CrCl < 40 mL/min) on 4.5 grams | 6.2 [2.3 to 10.6]
  Group 3 (CrCl < 40 mL/min) on 6.75 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40 mL/min) on 6.75 grams | 5.5 [5.1 to 5.8]
  Group 4 (HD) on 2.25 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 2.25 grams | 9.8 [9.8 to 9.8]
  Group 4 (HD) on 3.375 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 3.375 grams | 8.6 [8.6 to 8.6]
  Group 4 (HD) on 4.5 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 4.5 grams | 9.1 [9.1 to 9.1]
  Group 4 (HD) on 6.75 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 6.75 grams | 7.4 [6.5 to 8.4]

4. Secondary Outcome: Volume of Distribution of Piperacillin
Description: Volume of distribution (Vd) of piperacillin will be calculated from serum concentrations in both standard and high doses
Time Frame: 0, 1, 3, and 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: liters
Arm/Group | Standard Dose to High Dose Piperacillin/Tazobactam
Number analyzed (Participants) | 28
liters
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams: number analyzed (Participants) | 7
  Group 1 (CrCl >/= 80 mL/min) on 3.375 grams | 19.0 [14.1 to 24.7]
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 1 (CrCl >/= 80 mL/min) on 4.5 grams | 20.9 [13.6 to 27.6]
  Group 1 (CrCl >/= 80 mL/min) on 6.75 grams | 27.7 [14.9 to 61.0]
  Group 1 (CrCl >/= 80 mL/min) on 9 grams: number analyzed (Participants) | 3
  Group 1 (CrCl >/= 80 mL/min) on 9 grams | 20.1 [17.3 to 22.3]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 3.375 gram: number analyzed (Participants) | 6
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 3.375 gram | 31.6 [20.4 to 54.8]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 4.5 gram: number analyzed (Participants) | 2
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 4.5 gram | 20.3 [19.3 to 21.3]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 6.75 gram: number analyzed (Participants) | 7
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 6.75 gram | 31.7 [18.3 to 54.5]
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 9 gram: number analyzed (Participants) | 1
  Group 2 (CrCl >/= 40 to < 80 mL/min) on 9 gram | 48.8 [48.8 to 48.8]
  Group 3 (CrCl < 40mL/min) on 2.25 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40mL/min) on 2.25 grams | 22.9 [16.9 to 28.8]
  Group 3 (CrCl < 40mL/min) on 3.375 grams: number analyzed (Participants) | 1
  Group 3 (CrCl < 40mL/min) on 3.375 grams | 30.5 [30.5 to 30.5]
  Group 3 (CrCl < 40mL/min) on 4.5 grams: number analyzed (Participants) | 5
  Group 3 (CrCl < 40mL/min) on 4.5 grams | 26.3 [20.0 to 32.9]
  Group 3 (CrCl < 40mL/min) on 6.75 grams: number analyzed (Participants) | 2
  Group 3 (CrCl < 40mL/min) on 6.75 grams | 29.9 [23.5 to 36.3]
  Group 4 (HD) on 2.25 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 2.25 grams | 34.9 [34.9 to 34.9]
  Group 4 (HD) on 3.375 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 3.375 grams | 28.9 [28.9 to 28.9]
  Group 4 (HD) on 4.5 grams: number analyzed (Participants) | 1
  Group 4 (HD) on 4.5 grams | 24.6 [24.6 to 24.6]
  Group 4 (HD) on 6.75 grams: number analyzed (Participants) | 2
  Group 4 (HD) on 6.75 grams | 34.0 [29.7 to 38.3]

ADVERSE EVENTS:
Time Frame: Each patient was monitored daily for adverse reactions from study enrollment until two weeks after piperacillin-tazobactam was discontinued or until hospital discharge, whichever was sooner
Description: Pertinent lab values followed for signs of acute renal impairment, liver impairment, or hematologic abnormalities. Adverse reactions were promptly reported to the primary team and IRB. If study drug suspected to be responsible for an adverse reaction, the drug discontinued at the discretion of the primary care team. There were no deaths out of the 28 subjects at risk of death during study enrollment.
Arm/Group | Standard Dose to High Dose Piperacillin/Tazobactam
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 6/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose to High Dose Piperacillin/Tazobactam (N=29)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) — Nausea with one episode of vomiting, which resolved upon dose reduction in one patient on the 6.75 grams dose of piperacillin-tazobactam. Naranjo scale gave this a 6 as probably related to study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose to High Dose Piperacillin/Tazobactam (N=29)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) — Naranjo scale gave 2 patients a 2 and a 3 respectively, making adverse reaction possibly related to study drug. There were many confounders in these 2 patients regarding reasons for acute kidney injury.
Nausea (Gastrointestinal disorders) | 1 (1) — Mild in one patient that resolved while still on high dose of study drug. Naranjo scale gave this a 2 as possibly related to study drug
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Patient had cholecystitis and abdominal abscess. Symptoms subsided during treatment course with no dose adjustment. Naranjo scale gave this a 1 for possibly a study drug related event.
Diarrhea (Gastrointestinal disorders) | 1 (1) — one episode of loose stool after 4.5 gram dose which resolved spontaneously without dose adjustment. Naranjo scale gave this a 2, possibly related to study drug.
Delirium (Psychiatric disorders) | 1 (1) — one patient had acute onset delirium on high dose drug, biting off a few of his fingernails. Patient was also on lorazepam scheduled every 6 hours. Study drug dose reduced and lorazepam discontinued. Patient returned to baseline. Naranjo scale = 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No